CLINICAL TRIAL: NCT05195775
Title: Tadalafil as an Adjuvant to Therapy for Duchenne Muscular Dystrophy
Brief Title: Tadalafil as Adjuvant Therapy for DMD
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202102391; OCR41391 (Other: UF OnCore)
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: therapy; treatment strategy; vasodilator; exercise
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Motor Activity | interventions — Tadalafil

STUDY DESIGN:
Intervention Model Description: Pre/post single dose tadalafil
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tadalafil plus BOLD-MRI (Schedule A) (Experimental): The intervention is the same as in Schedule B; this arm will use BOLD-MRI as the technique to monitor drug impact on skeletal muscle.
  Interventions: Drug: Tadalafil
- Tadalafil plus Doppler ultrasound (Schedule B) (Experimental): The intervention is the same as in Schedule A; this arm will use Doppler ultrasound as the technique to monitor drug impact on skeletal muscle.
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — Patient will be randomized to one dose of 0.6 mg/kg tadalafill on one of two study visits. On both visits, assessments (MRI, exercise testing, clinical function) will be performed 3 hours after time of dosing.
  Other Names: Cialis
  Arms: Tadalafil plus BOLD-MRI (Schedule A)
Drug: Tadalafil — Patient will be randomized to one dose of 0.6 mg/kg tadalafill on one of two study visits. On both visits, assessments (Doppler US, exercise testing, clinical function) will be performed 3 hours after time of dosing.
  Other Names: Cialis
  Arms: Tadalafil plus Doppler ultrasound (Schedule B)

SUMMARY:
This project will assess the vascular responsiveness in leg muscles of boys with Duchenne muscular dystrophy (DMD) to one single dose of tadalafil, a common vasodilator drug, using non-invasive techniques (MRI or Doppler ultrasound) and exercise testing. These findings will provide proof of concept for a subsequent intervention study to demonstrate efficacy of longer-term tadalafil to counter sympathetic vasoconstriction and slow disease progression in DMD. It will also inform whether a group of patients do not respond to the drug.

DETAILED DESCRIPTION:
This project will target up to 25 ambulatory boys with DMD aged 7-13 years. Because the vascular impact of tadalafil is immediate, we will confirm that the drug target is valid target in lower extremities by assessing the change in post-exercise microvascular perfusion using Blood Oxygen Level-Dependent (BOLD) MRI or change in post-exercise hyperemia using Doppler ultrasonography. We will also assess the functional impact of the drug through exercise testing. Patients will be randomized to undergo the above-mentioned assessments with or without the study drug on two separate visits. Time function tests, MRI-based fat fraction and inflammation measurements will also be obtained in all patients, thus characterizing disease severity and provide a sampling of information on whether a subset of patients do not respond to the drug. This information may be used to inform future trials as to the appropriate target population for PDE5i as well as account for potential failures in a previously published phase 3 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DMD confirmed by 1) clinical history with features before the age of five, 2) physical examination, 3) elevated serum creatine kinase level and 4) absence of dystrophin expression, as determined by immunostaining or Western blot (<2%) and/or DNA confirmation of dystrophin mutation.
* Minimum entry age of 7.0 years
* Ambulatory

Exclusion Criteria:

* Older than 13.0 years of age
* Contraindication to an MR examination (e.g. aneurysm clip, severe claustrophobia, magnetic implants)
* Presence of unstable medical problems
* Presence of a secondary condition that impacts muscle function or muscle metabolism (e.g. myasthenia gravis, endocrine disorder, mitochondrial disease)
* Contraindications to Tadalafil (use of nitrates, alpha-adrenergic blockers, other PDE5A inhibitors)

Ages: 7 Years to 13 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Duchenne Muscular Dystrophy is an X-linked disorder, and therefore predominantly in males. As a result, we are limiting our children study participants to males.
Enrollment: 25 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2025-09-05 (Estimated); Study Completion 2025-09-05 (Estimated)

PRIMARY OUTCOMES:
Change in post-contractile BOLD response after tadalafil dosing | MRI will be done 3 hours after dosing/no-dosing on two separate study visits
  MRI technique to measure microvascular function in skeletal muscle
Change in post-exercise hyperemia after tadalafil dosing | Doppler ultrasound will be done 3 hours after dosing/no-dosing on two separate study visits
  Doppler ultrasound will be used to measure blood flow

SECONDARY OUTCOMES:
Change in submaximal exercise capacity after tadalafil dosing | Cycle testing will be done 4 hours after dosing/no-dosing on two separate study visits
  incremental cardiopulmonary exercise testing on cycle ergometer will be performed to measure heart rate and parameters of exercise performance.

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Taivassalo, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No